CLINICAL TRIAL: NCT02512419
Title: Developing a Text-Message Enhanced Physical Activity Intervention for Latino Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dr.Bess Marcus, Professor and Chair, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Activo R21; R21NR014911 (NIH)
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Inactivity
Keywords: Physical Activity; Latinos; Mexican American Men; Spanish-Language; Text-Message
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text-Enhanced Physical Activity Intervention Arm (Experimental): The Spanish-language PA intervention is based on Social Cognitive Theory (SCT) and Transtheoretical Model (TTM), and emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting physical activity goals).
  Interventions: Behavioral: Text-Enhanced Physical Activity Intervention Arm; Device: Actigraph GT3X
- Health Education Control Arm (Active Comparator): The health education control arm will receive the publicly available NHBLI Spanish-language booklets on heart-healthy behaviors for Latinos, which include information on PA, diet, and stress management.
  Interventions: Behavioral: Health Education Control Arm; Device: Actigraph GT3X

INTERVENTIONS:
Behavioral: Text-Enhanced Physical Activity Intervention Arm — Participants in the Text-Enhanced Physical Activity intervention arm of the study receive a Spanish language, motivationally-tailored, print-based + text-message physical activity intervention that specifically addresses the physical activity barriers and intervention needs/preferences of Mexican and Mexican American men.
  Arms: Text-Enhanced Physical Activity Intervention Arm
Behavioral: Health Education Control Arm — Participants will receive a Spanish language, print-based Wellness Contact control intervention addressing relevant health topics other than physical activity.
  Arms: Health Education Control Arm
Device: Actigraph GT3X

SUMMARY:
The aim of this study is to build upon our tailored print intervention by developing new text-delivered intervention materials to complement our print-based physical activity (PA) intervention. In Phase 1 we will conduct 6 focus groups with Mexican and Mexican American (MA) men to determine content, frequency, and types of text messages desired, and to identify cultural themes to incorporate into existing and new materials. Themes from the focus groups and sample text messages will be presented to a confirmatory focus group panel. Phase 2 will be a 6-month pilot randomized controlled trial with Mexican and MA men (N=60) to test the text-enhanced, Spanish language, individually tailored PA intervention vs. publicly available, Spanish language health education materials, including information on PA, diet, and stress management. This will be followed by post-intervention qualitative interviews to solicit suggestions for improvements to help further refine the program. The proposed pilot will support a future R01 to establish the efficacy of this multi-media, multi-level PA intervention for Mexican and MA men.

DETAILED DESCRIPTION:
The proposed research addresses serious public health concerns (inactivity, health disparities) in a large, rapidly growing population of Mexican American (MA) men who are markedly less physically active than men of other ethnicities and suffer from higher prevalence of conditions related to sedentary lifestyle. While this population is clearly in need of physical activity (PA) interventions, to date none have specifically targeted MA men. In fact, the majority of PA interventions for Latinos have exclusively included women and/or are designed around female preferences.The proposed study will address the needs and barriers to PA in MA men by developing text message-delivered intervention materials based on Social Cognitive Theory (SCT) to complement an individually tailored, theory-based print material PA intervention for Spanish speaking Mexican and MA men. Text messaging could be a particularly effective and appealing channel for increasing PA in this target population as it allows for participant interaction, real-time accountability, and immediate feedback, features which MA men in the demonstration trial of our print intervention specifically requested. Text-based interventions have been shown to improve a number of health behaviors, including PA. A recent review of texting interventions found that they were generally well received and effective in reducing inactivity, weight, and waist circumference,5 and a meta-analysis found a moderate effect size (g = 0.54) for using mobile devices to increase PA. However, few of these trials targeted underserved populations, and none specifically targeted Latinos. Cell phone ownership is high in Latino adults (86% vs. 84% in non-Latino Whites), and Latinos are actually the most likely to use mobile phones for text messaging, with 85% reporting regularly sending and receiving texts (compared to 79% of Whites). Thus this is a familiar, convenient channel for delivering new intervention materials. Additionally, as Latinos also face environmental barriers to PA, in the current proposal we will enhance the individually tailored psychosocial print-based materials by developing materials targeting barriers in home and work environments. This multi-media, multi-level approach has potential for broad reach at relatively low cost, which could help reduce health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Generally healthy (If asthma, controlled high blood pressure and/or controlled type II diabetes, may be able to participate with physician consent)
* Sedentary (Less than 60 minutes per week of moderate or vigorous physical activity)
* Mexican and/or Mexican American (self-identified)
* Must be able to read and write Spanish fluently
* 18 - 65 years of age
* Planning on living in the area for the next 6 months
* Own a cell phone capable of sending and receiving text messages

Exclusion Criteria:

* Body Mass Index(BMI) greater than 45
* Not able to walk continuously for 30 minutes/limited ability to complete daily activity or ability to exercise
* Exercise is against advice of doctor
* Heart disease/treatment
* Heart murmur
* Angina/chest pain or Angina/chest pain with exertion
* Palpitations
* Stroke/Transient Ischemic Attacks
* Peripheral Vascular Disease
* Type I Diabetes
* Uncontrolled Type II Diabetes
* Chronic Infectious Disease - HIV, Hepatitis
* Chronic liver disease
* Cystic Fibrosis
* Abnormal EKG on last EKG performed
* Emphysema, Chronic bronchitis, Chronic Obstructive Pulmonary Disease
* Seizure in past year
* Surgery in past year on heart, lung, joint, orthopedic surgery
* Surgery pending in next year on lung, joint, orthopedic surgery
* Unusual/concerning shortness of breath
* Asthma (may be able to participate with physician consent)
* High blood pressure/high blood pressure medication (may be able to participate with physician consent)
* Use of beta blockers
* Abnormal Medical Stress Test
* Musculoskeletal problems
* Fainting/dizziness more than 3 times in past year OR interferes with daily activities OR causes loss of balance
* Cancer treatment in past 3 months
* Hospitalized for psychiatric disorder in past 3 years or suicidal

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07; Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Larsen BA, Benitez TJ, Mendoza-Vasconez AS, Hartman SJ, Linke SE, Pekmezi DJ, Dunsiger SI, Nodora JN, Gans KM, Marcus BH. Randomized Trial of a Physical Activity Intervention for Latino Men: Activo. Am J Prev Med. 2020 Aug;59(2):219-227. doi: 10.1016/j.amepre.2020.03.007. Epub 2020 May 21. PMID 32448552

RESULTS

PARTICIPANT FLOW:
Groups:
- Text-Enhanced Physical Activity Intervention Arm: The Spanish-language PA intervention is based on SCT and Transtheoretical Model (TTM), and emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting PA goals).
  Text-Enhanced Physical Activity Intervention Arm: Participants in the Text-Enhanced Physical Activity intervention arm of the study receive a Spanish language, motivationally-tailored, print-based + text-message physical activity intervention that specifically addresses the physical activity barriers and intervention needs/preferences of Mexican and Mexican American men.
  Actigraph GT3X
- Health Education Control Arm: The health education control arm will receive the publicly available NHBLI Spanish-language booklets on heart-healthy behaviors for Latinos, which include information on PA, diet, and stress management.
  Health Education Control Arm: Participants will receive a Spanish language, print-based Wellness Contact control intervention addressing relevant health topics other than physical activity.
  Actigraph GT3X
Period: Overall Study
Arm/Group | Text-Enhanced Physical Activity Intervention Arm | Health Education Control Arm
Started | 24 | 24
Completed | 22 (2 participants became ineligible after enrolling therefore were not included in analysis.) | 24
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Two participants were randomized never started and thus removed from subsequent analyses.
Groups:
- Text-Enhanced Physical Activity Intervention Arm: The Spanish-language Physical Activity intervention is based on Social Cognitive Theory (SCT) and Transtheoretical Model (TTM), and emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting physical activity goals).
  Text-Enhanced Physical Activity Intervention Arm: Participants in the Text-Enhanced Physical Activity intervention arm of the study receive a Spanish language, motivationally-tailored, print-based + text-message physical activity intervention that specifically addresses the physical activity barriers and intervention needs/preferences of Mexican and Mexican American men.
  Actigraph GT3X
- Total: Total of all reporting groups
Arm/Group | Text-Enhanced Physical Activity Intervention Arm | Health Education Control Arm | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.23 (10.34) | 41.96 (11.07) | 43.04 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 24 | 46
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46
Objectively Measured Physical Activity [Median (Inter-Quartile Range); unit: minutes/week] — Baseline objectively measured physical activity of at least moderate intensity (MVPA) collected via accelerometer
  minutes/week | 10 [0 to 42.5] | 21 [0 to 59] | 10.5 [0 to 49.25]
Self-Reported Physical Activity [Median (Inter-Quartile Range); unit: minutes/week] — Subjectively reported baseline minutes of at least moderate intensity physical activity (MVPA) as reported on the 7 day physical activity recall (PAR)
  minutes/week | 10 [0 to 45] | 5 [0 to 43.75] | 10 [0 to 42.5]

OUTCOME MEASURES:

1. Primary Outcome: Objectively Measured Physical Activity of at Least Moderate Intensity (MVPA) by the Actigraph GT3X+
Description: Participants will wear an Actigraph GT3X+ accelerometer, which measures movement and intensity of activity and has been validated against heart rate telemetry and total energy expenditure.
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: minutes/week
Arm/Group | Text-Enhanced Physical Activity Intervention Arm | Health Education Control Arm
Number analyzed (Participants) | 22 | 24
minutes/week
  Baseline | 10 [0 to 42.5] | 21 [0 to 59]
  6 Months | 57.5 [18.5 to 104.5] | 23 [0 to 76.25]
Statistical Analysis 1: Comparison: Text-Enhanced Physical Activity Intervention Arm vs Health Education Control Arm; To examine potential intervention effects on the primary outcome (MVPA at 6 months), we used a series of quantile regression models which model median outcome at follow-up as a function of baseline value of the outcome (MVPA), treatment condition and covariates. Note that the adjusted difference in median MVPA between conditions at follow-up will not equal the difference in median minutes as seen in the unadjusted tables as these estimates are adjusted; Test type: Superiority; p = .04, quantile regression; Models regressed outcome at 6 months on treatment assigned, baseline value of the outcome and actigraph wear time. Effect sizes reported are adjusted; regression parameter (median diff) = 37.52, Standard Error of Mean 18.01 — Effects are unstandardized regression coefficients. They represent difference in median outcome between conditions at 6m controlling for baseline and covariates

2. Primary Outcome: Self Reported Min/Week of MVPA
Description: Self reported physical activity (collected via 7 day PAR)
Time Frame: baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: min/week
Arm/Group | Text-Enhanced Physical Activity Intervention Arm | Health Education Control Arm
Number analyzed (Participants) | 22 | 24
min/week
  Baseline | 10 [0 to 45] | 5 [0 to 43.75]
  6 Months | 95 [15 to 180] | 52.5 [16.25 to 298.50]
Statistical Analysis 1: Comparison: Text-Enhanced Physical Activity Intervention Arm vs Health Education Control Arm; Quantile regression was used; Test type: Superiority; p = 0.10, quantile regression; Median Difference (Final Values) = 42.36, Standard Error of Mean 38.83

ADVERSE EVENTS:
Time Frame: 28 months (first baseline visit to last 6 month visit)
Arm/Group | Text-Enhanced Physical Activity Intervention Arm | Health Education Control Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT02512419/Prot_SAP_000.pdf